CLINICAL TRIAL: NCT02136706
Title: Feasibility and Diagnostic Accuracy of Myocardial SPECT Using Early Imaging Protocol: A Pilot Study
Brief Title: Feasibility and Diagnostic Accuracy of Myocardial SPECT Using Early Imaging Protocol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor and site were unable to complete a final contract to support the study
Sponsor: Medhat Osman MD (U.S. Federal Agency)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Medhat Osman MD, Professor of Radiology, Director of Nuclear Medicine and Pet/CT, VA St. Louis Health Care System
Organization: VA St. Louis Health Care System (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REGA-14A01
Record Dates: First submitted 2014-05-04; First posted 2014-05-13 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Stable coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 10/30 min rest/stress (No Intervention): Rest and stress T99m-MPI obtained 10 minutes and 30 minutes after tracer injection. After the myocardial perfusion imaging the investigators will have 10 minute waiting period to take images and then wait the 30 minutes, standard of care to take the images.
  Interventions: Procedure: Myocardial Perfusion imaging with 10 minute waiting period

INTERVENTIONS:
Procedure: Myocardial Perfusion imaging with 10 minute waiting period — After the Myocardial Perfusion Imaging testing the investigators will wait 10 minutes to take images and then wait the 30 minute standard of care time to take images.

SUMMARY:
Encouraged by the recent data published ,the investigators think that a waiting time of 10 minutes is feasible while preserving diagnostic accuracy and would like to assess the feasibility and diagnostic efficacy of W10 compared with W30 imaging in a pilot study. By combining W10 imaging with half-time acquisition, the time of the technetium-99m myocardial perfusion imaging procedure could be shortened by at least 50%, lasting only 40 minutes for W10 (10-minute waiting) imaging compared with 90 minutes for W30 imaging (30-minute waiting).

The investigators hypothesize that (1) W10 MPI is clinically feasible and tolerable by the patients, that (2) W10 MPI provides high image quality and that (3) W10 MPI provides diagnostic accuracy comparable to W30 MPI.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 and ≤ 89 years of age of any race /ethnicity
* Patient has undergone or is being scheduled for a clinically indicated CardiacCath with or without angioplasty
* Patient may have suffered myocardial infarction more than 3 days before T99m-MPI
* Patient may have undergone percutaneous transluminal coronary angioplasty (PTCA) or coronary stent placement more than 3 days prior to T99m-Myocardial Perfusion Imaging (MPI)
* Interval between T99m-MPI and CardiacCath is within 30 days
* Females cannot be pregnant or lactating
* Women of no child-bearing potential (post-menopausal defined as amenorrhea ≥ 12 consecutive months, or because they have undergone successful surgical sterilization and deny current history of pregnancy and nursing). These subjects do not require serum pregnancy test on the day of the study
* Women of childbearing potential will require a negative serum pregnancy test, performed on the day of the study
* Provide signed Informed Consent prior to undergoing the study procedures

Exclusion Criteria:

* Patients less than 18 and ≥89 years of age
* Patient has been involved in any other investigative, radioactive research procedure within 7 days and during the study participation period
* History of 2nd or 3rd degree Atrio-ventricular-block, or sinus node dysfunction unless the patients have a functioning artificial pacemaker
* Current ventricular tachycardia, atrial fibrillation, atrial tachycardia, or atrial flutter
* Current unstable angina or cardiovascular instability
* Current history of exacerbated Chronic Obstructive Pulmonary Disease (COPD) or asthma
* Known hypersensitivity or contraindication to regadenoson or aminophylline
* Use of caffeinated substance, dipyridamole-containing medication, aminophylline, or xanthines containing medication (e.g. theophylline) within the 12 hours prior to Lexiscan administration

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Visual and semi-quantitative evaluation of W10 and W30 studies. | Day 1of testing
  The investigators will evaluate image quality of W10 and W30-qualitatively (visually) by 2 independent readers and semi-qualitatively by means of region of interest (ROI) count/pixels parameters of W10 and W30 data and compare their diagnostic accuracy for the diagnosis of myocardial ischemia and infarction.

SECONDARY OUTCOMES:
Tolerability Questionnaire | Day 1 of testing
  Each patient will complete a total of 6 questionnaires on the day of testing before and after each stress W10 and W30 scanning. The participants will be asked to rate how they felt, and if present, how they perceived their headache during scanning. Patients will also be asked how they felt and how severe was their headache when comparing the rest W10 and W30 and the stress W10 and W30.
Feasibility of W10 by written documentation. | Day 1 of testing
  By documenting any technical or clinical difficulties during the W10 procedure

IPD SHARING:
Plan to Share IPD: No